CLINICAL TRIAL: NCT02340611
Title: A Proof of Concept Clinical Trial of the Combination Cediranib-Olaparib at the Time of Disease Progression on Olaparib in Ovarian Cancer
Brief Title: A Study of Cediranib and Olaparib at the Time Ovarian Cancer Worsens on Olaparib
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: e-Volve
Record Dates: First submitted 2015-01-13; First posted 2015-01-16 (Estimated); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — olaparib; cediranib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cediranib and Olaparib (Experimental): Cediranib, 20 mg , orally, once a day, every day. Olaparib, 150 mg or 200 mg (depending on previous treatment dose), orally, once a day, every day.
  Interventions: Drug: Olaparib; Drug: Cediranib

INTERVENTIONS:
Drug: Olaparib — Polyadenosine 5'diphosphoribose polymerase (PARP) Inhibitor
  Other Names: AZD2281; KU-0059436
Drug: Cediranib — Vascular endothelial growth factor (VEGF) receptor tyrosine kinase inhibitor that is a potent inhibitor of all three VEGF receptors (VEGFR-1, -2 and -3)
  Other Names: AZD2171; Recentin™

SUMMARY:
This is a phase 2 study (the second phase in testing a new drug or drug combination) to see how useful adding investigational drug cediranib to olaparib after disease progression on olaparib alone in patients with ovarian cancer.

DETAILED DESCRIPTION:
Cediranib works by blocking (inhibiting) several specific proteins in cancer cells called the vascular endothelial growth factor (VEGF) receptors. These proteins are important in the formation of blood vessels to the tumor. It is believed that many tumors survive because the blood vessels on the tumors bring oxygen and nutrients to the cancer cells which enable them to grow. If the formation of the blood vessels is blocked, the tumor cells may die.

Olaparib works by blocking protein called poly [adenosine diphosphate-ribose] polymerase (PARP). PARP is an important protein which tries to fix damaged deoxyribonucleic acid (DNA, molecules that contain important instructions for the development of cells). Many cancers are though develop from damaged DNA. By blocking PARP from fixing damaged DNA, the tumor cells may die.

Adding cediranib to olaparib, and therefore blocking several different mechanisms for cancer growth, may stop tumor growth.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Performance status 2 or less
* Ovarian cancer, high grade serous or high grade endometrioid histology subtype
* Radiographically documented disease progression per RECIST 1.1
* Progression on olaparib therapy after an initial good response (more than 6 months)
* Patients must have adequate bone marrow, renal and hepatic function per local laboratory reference range
* Ongoing prior toxicities related to previous treatments recovered to grade 2 or less
* LVEF>50% by echocardiograms or MUGA
* Urine dipstick for proteinuria <2+
* Willing to undergo tumour biopsy pre-treatment
* Life expectancy of greater than 3 months
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Current bowel obstruction
* Known brain metastases
* Mean QTc >470 msec (with Bazett's correction) in screening ECG or history of familial long QT syndrome.
* Uncontrolled intercurrent illness including, but not limited to hypertension, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* A New York Heart Association classification of III or IV requiring concurrent use of drugs or biologics with proarrhythmic potential.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to olaparib or cediranib
* Unable to swallow orally administered medication and/or gastrointestinal disorders likely to interfere with absorption of the study medication.
* Myelodysplastic syndrome/acute myeloid leukaemia
* Immuno-compromised patients, e.g., patients who are known to be serologically positive for human immunodeficiency virus (HIV), patients with known active hepatitis (i.e.,hepatitis B or C) due to risk of transmitting the infection through blood or other body fluids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-06; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Percentage of patients whose cancer shrinks or disappears after treatment | 2 years

SECONDARY OUTCOMES:
Percentage of decrease in CA-125 levels after treatment | 2 years
Mutation status of genes compared to response to treatment | 2 years
Number of occurences per side effect and severity | 2 years
Assess patient reported outcomes during treatment | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Amit Oza, M.D., Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada